CLINICAL TRIAL: NCT02841631
Title: Investigation Into the Infectivity Levels of Human Papilloma Virus (HPV) in Tonsillar Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Derby (Other)
Responsible Party: Principal Investigator, Raguwinder Sahota, Associate Lecturer, University of Derby
Other Study IDs: IRAS 194857
Record Dates: First submitted 2016-07-15; First posted 2016-07-22 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Human Papillomavirus, Palatine Tonsil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral rinse and Tonsillectomy specimens
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Post-Tonsillectomy: Subjects undergoing tonsillectomy for non-cancer reasons including operations for: recurrent tonsillitis, asymmetric tonsils, snoring surgery or obstructive sleep apnoea.
  Interventions: Genetic: HPV status and typing of tissue

INTERVENTIONS:
Genetic: HPV status and typing of tissue — HPV status and typing of tissue

SUMMARY:
Human Papilloma Virus (HPV) has been shown to be a cause of Head & Neck Squamous Cell Carcinoma (HNSCC) and the majority of current studies focus on what is happening in patients with a HPV HNSCC. But there is limited investigation into HPV infection in the oropharynx of patients who do not have HNSCC. The current incidence of oral HPV infection is not known in the general population locally and there is also limited information on what particular localities within the mouth that patients' harbour HPV infection what strains are present and if there are any differences in viral load.

Therefore the aim of this project is to investigate within patients that undergo tonsillectomies the rate of HPV infection in tonsils to determine the amount of HPV present within the community.

DETAILED DESCRIPTION:
Patients are having no additional invasive testing than is all ready being carried out for their care pertaining to their tonsillar tissue. Patients are routinely swabbed pre-operative for evidence of MRSA, this trial would add an extra swabbing procedure for the mouth.

The ethical implications are related to the tissue which is being tested for a virus that can be implicated in head and neck squamous cancer. These patients would not normally be aware of HPV infection and this would raise an new health burden in these patient who are likely to be fit and well. The research team would be suitable to counsel patients from any worries related to HPV infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing routine tonsillectomies who can provide consent to participate over the age of 18 years old would eligible to enter the study. They would all ready be listed for a tonsillectomy after being seen by an ENT surgeon.

Exclusion Criteria:

* Patients unable to give informed consent
* If the tonsillectomy is carried out to diagnose cancer
* Patient chooses to decline recruitment into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a routine tonsillectomy operation for non-cancerous reasons at the hospital will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Rate of oral and tonsillar HPV infection in patients undergoing tonsillectomies and to investigate any links with lifestyle. | over the 3 years of the study
  The aim of this project is to examine the rate of oral and tonsillar HPV infection in patients undergoing tonsillectomies and to investigate any links with lifestyle.

SECONDARY OUTCOMES:
Validation of a reproducible oral HPV screening method to detect HPV from saliva samples and also tonsillar tissue to investigate rates of oral HPV infection. | over the 3 years of the study
  Validation of a reproducible oral HPV screening method to detect HPV from saliva samples and also tonsillar tissue to investigate rates of oral HPV infection. The investigators will be using quantitative PCR to detect the strains of HPV and the viral load.
Quantification and typing via quantitative PCR of detectable HPV infection from saliva and tonsillar samples to investigate any differences between samples from the same patient and also different patients. | over the 3 years of the study
  Quantification and typing of detectable HPV infection from saliva and tonsillar samples to investigate any differences between samples from the same patient and also different patients.
Examination of viral load and also expression levels of the HPV viral oncogenes (E6 and E7) from infected tissue to investigate any differences in protein expression between different patients. | over the 3 years of the study
  Examination of viral load and also expression levels of the HPV viral oncogenes, E6 and E7, from infected tissue to investigate any differences in protein expression between different patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Derby Hospital, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided